CLINICAL TRIAL: NCT03637439
Title: Effects of Ultrasound-guided Percutaneous Neuromodulation on Flexibility and Hamstring Force
Brief Title: Neuromodulation in Patients With Hamstring Shortening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Antonio Garcia Vidal (Other)
Collaborators: Universidad de Murcia (Other)
Responsible Party: Sponsor-Investigator, Jose Antonio Garcia Vidal, Physiotherapist, PhD, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1858/2018
Record Dates: First submitted 2018-08-11; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Hamstring Contractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNM group (Experimental): Subjects were treated only once. Specifically, this consisted in the application of a square wave biphasic electrical current, with 10 Hz frequency, a 250µs pulse width, and the maximal tolerable intensity to cause an exacerbated muscle contraction for a total of 1.5 mins, according to the protocol (Valera & Minaya). The subjects were lying prone in decubitus. The middle part of the sciatic nerve was located using an ultrasound machine (cross section), then an acupuncture needle (0.30 mm x 40 mm) was inserted in a short axis approach, perpendicular to the surface of the skin, to the perineurium of the sciatic nerve.
  Interventions: Other: Ultrasound-guided Percutaneous Neuromodulation
- Control group (Sham Comparator): The subjects were lying prone in decubitus. The same puncture protocol was performed on the sciatic nerve for 1.5 minutes, but without the application of electricity.
  Interventions: Other: Ultrasound-guided Percutaneous Needle

INTERVENTIONS:
Other: Ultrasound-guided Percutaneous Neuromodulation — It's a new intervention of sport physiotherapy. It´s an invasive technique. It is necessary an ultrasound
  Arms: PNM group
Other: Ultrasound-guided Percutaneous Needle — Same protocol without electricity
  Arms: Control group

SUMMARY:
The flexibility of the hamstrings is a very important component both for general health and when exercising. The lack of hamstring flexibility has been related to the increase in the likelihood of suffering a large number of musculoskeletal pathologies, due to the possibility of causing important muscle imbalances, which include lumbar spine pathologies, such as disc hernias or spondyloarthrosis. In addition, the decrease in the flexibility of the hamstring musculature is also related to the increased likelihood of suffering muscle strains, patellar tendon tendinopathies, femoropatellar syndrome and decreased lumbopelvic rhythm.

Clinically, an invasive technique has appeared, known as Ultrasound-guided Percutaneous Neuromodulation (PNM). This minimally invasive intervention consists in the application of a percutaneous electrical stimulation (PES) through an acupuncture needle-like electrode that is placed in close proximity to the nerve or motor point of the muscle with ultrasound guidance. At the clinical level, the PES is always used with the therapeutic aim of relieving chronic pain and neuropathic pain. Similarly, in sports, PES is used with the aim of improving muscular activity. Therefore, according to the characteristics and the therapeutic benefits of this technique, further research is needed to discover multiple clinical indications.

The aim of this study was to examine the effects on flexibility and strength of an ultrasound-guided percutaneous neuromodulation intervention in patients with shortening of the hamstring muscles.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* to practice some sports activity 2 or more times a week
* get less than 70º in PKE (Passive Knee Extension) with hip 90º

Exclusion Criteria:

* any previous surgery or acute trauma in the back or lower extremity.
* pain at the time of performing the assessment tests
* belonephobia
* anticoagulant consumption
* pregnancy
* hemorrhagic disorders
* immunosuppression
* inability to understand or carry out evaluations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
Change from Passive Knee Extension 90º [PKE 90º] [Hamstring Flexibility test] 5 minutes after intervention | Baseline and 5 minutes after intervention
  Passive Knee Extension with hip 90º. The examiner will measure the popliteal angle (between the femur and the tibia) with a goniometer.

SECONDARY OUTCOMES:
Change from Sit and Reach Flexibility Test [Hamstring Flexibility test] 5 minutes after intervention | Baseline and 5 minutes after intervention
  The sit and reach test is a common measure of flexibility of the lower back and hamstring muscles. Using a standard sit and reach box, the participant sat on the floor with shoes on, and fully extended one leg so that the sole of the foot was flat against the end of the box. She then extended her arms forward, placing one hand on top of the other. With palms down, she reached forward sling hands along the measuring scale as far as possible without bending the knee of the extended leg.
Change from Stand and Reach Flexibility Test [Hamstring Flexibility test] 5 minutes after intervention | Baseline and 5 minutes after intervention
  The volunteer standing with his knees extended tries to touch the ground with his extended hands. The examiner will measure with a ruler the distance in centimeters between the floor and the tips of fingers.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy Department. University of Murcia, Murcia, Spain